CLINICAL TRIAL: NCT00532337
Title: A Multi-centre, Randomized, Double Blind, Parallel Group Study to Investigate Efficacy and Safety of ONO-5334 in Postmenopausal Women With Osteopenia or Osteoporosis
Brief Title: Controlled Study of ONO-5334 in Postmenopausal Women With Osteopenia or Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5334POE003
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Osteoporosis; Osteopenia
Keywords: ONO-5334; osteoporosis; osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — ONO-5334

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- P (Placebo Comparator)
  Interventions: Drug: ONO-5334
- E1 (Experimental)
  Interventions: Drug: ONO-5334
- E2 (Experimental)
  Interventions: Drug: ONO-5334
- E3 (Experimental)
  Interventions: Drug: ONO-5334
- A (Active Comparator)
  Interventions: Drug: ONO-5334

INTERVENTIONS:
Drug: ONO-5334 — Placebo - 24/mos.
  Arms: P
Drug: ONO-5334 — 100mg QD /24 months
  Arms: E1
Drug: ONO-5334 — 50mg BID /24 mos.
  Arms: E2
Drug: ONO-5334 — 300mg QD /24 mos.
  Arms: E3
Drug: ONO-5334 — Alendronate 70mg once weekly / 24 mos
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-5334 in postmenopausal women with osteopenia or osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoporosis defined as a value DXA BMD 2.5 SD or more below the young adult mean (T-score, ≤-2.5) at the lumbar spine (L1 to L4) or total hip, OR

* Osteoporosis defined as a value of DXA BMD more than 1 SD below the young adult mean, but less than 2.5 SD below this value (T-score <-1 and >2.5) at the lumbar spine (L1 to L4) or total hip.

Exclusion Criteria:

1. Patients with a value of DXA BMD more that 3.5 SD below the young adult mean, (T-score <-3.5) at the lumbar spine (L1 to L4) or total hip.
2. Osteoporosis patients (T-score ≤-2.5) who have any vertebral fragility fracture between T4 and L4 inclusive.
3. Osteopenia patients (T-score <-1 and >-2.5) who have no vertebral fragility fractures between T4 and L4 inclusive, OR

   * Osteopenia patients (T-score <-1 and >-2.5) who have two or more vertebral fragility fractures between T4 and L4 inclusive.
4. Patients who have abnormalities of the lumbar spine or femoral neck or internal organs around them precluding the assessment of BMD.
5. Patients who have secondary causes of osteoporosis or other disorders of bone and mineral metabolism.
6. Other exclusion criteria as specified in the study protocol.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mean bone mineral density of the lumbar spine (L 1-4 BMD) | 12 months

SECONDARY OUTCOMES:
Bone mineral density at hip, Biochemical markers of bone turnover | during course of treatment of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Kuwayama, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Andromed Noord Groningen, Damsterdiep 9, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Eastell R, Nagase S, Small M, Boonen S, Spector T, Ohyama M, Kuwayama T, Deacon S. Effect of ONO-5334 on bone mineral density and biochemical markers of bone turnover in postmenopausal osteoporosis: 2-year results from the OCEAN study. J Bone Miner Res. 2014 Feb;29(2):458-66. doi: 10.1002/jbmr.2047. PMID 23873670